CLINICAL TRIAL: NCT03906448
Title: A Phase 2, Historically Controlled Study Testing the Efficacy of TTFields (Optune®) With Adjuvant Temozolomide in High Risk WHO Grade II and III Astrocytomas (FORWARD)
Brief Title: FORWARD Optune and Adjuvant TMZ in Grade II/III Astrocytoma
Acronym: FORWARD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated because the Study Chair/IDE Sponsor and Novocure determined that conducting this trial was not feasible without CMS approval.
Sponsor: University of Florida (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201800600; OCR17711 (Other: UF OnCore)
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Astrocytoma, Grade II; Astrocytoma, Grade III
MeSH Terms: conditions — Astrocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Astrocytoma Patients (Experimental): Patients newly diagnosed with Grade II and III astrocytoma.
  Interventions: Combination Product: TTFields with adjuvant temozolomide
- Control Arm (No Intervention): Data collection from medical record only

INTERVENTIONS:
Combination Product: TTFields with adjuvant temozolomide — Patients will begin study treatment with temozolomide and TTFields within 2 weeks of the baseline evaluation, and no later than 6 weeks from last dose of concomitant temozolomide or radiation therapy (the latter of the two). A minimum of 6 and a maximum of 12 cycles of adjuvant temozolomide will be given, depending on tolerability and toxicity.
  Other Names: Optune
  Arms: Astrocytoma Patients

SUMMARY:
This is a phase 2, multi-institutional, historically-controlled, study of 100 patients with newly diagnosed Grade II and III astrocytoma comparing the combination of TTFields with adjuvant temozolomide versus temozolomide alone in historical controls after the completion of definitive chemoradiotherapy. Study treatment may continue past first tumor recurrence. The primary endpoint will be overall survival.

DETAILED DESCRIPTION:
Patients with newly diagnosed high-risk Grade II or III astrocytoma must undergo maximal safe resection (biopsy alone may be eligible) and chemoradiotherapy: concomitant 75mg/m2 daily temozolomide with 80% prescribed dose completed and RT with minimal RT dose of 40 Gy delivered.

Within three weeks prior to beginning adjuvant temozolomide, all patients will undergo a Baseline contrast-enhanced MRI of the brain. Within two weeks prior to beginning adjuvant temozolomide, all patients will undergo baseline assessments. Patients will begin study treatment with temozolomide and TTFields within 2 weeks of the baseline evaluation, and no later than 6 weeks from last dose of concomitant temozolomide or radiation therapy (the latter of the two). A minimum of 6 and a maximum of 12 cycles of adjuvant temozolomide will be given. Patients will be seen and examined before each cycle of temozolomide. After a maximum of 12 cycles of adjuvant temozolomide, patients will be seen every 8 weeks. Brain MRI and QoL assessments will be performed every 8 weeks following the baseline MRI for the first 2 years then every 3 months thereafter until second progression (when TTFields treatment will be terminated).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Life expectancy of at least 3 months
* Histologic confirmation of WHO Grade II or III astrocytoma---mixed oligoastrocytomas are permitted
* 1p/19q intact per FISH and/or ATRX mutation(s) per immunohistochemistry or next-generation sequencing (e.g. Foundation Medicine, TEMPUS, Caris, or similar CLIA-certified sequencing service)
* Mutational identity determined by CLIA-certified sequencing including:

  1. IDH1/2 wildtype (i.e. lack of detectable mutations on the sequencing report) and
  2. TERT promoter mutation
* Karnofsky performance status ≥70%
* Maximal safe resection---biopsy alone is allowed
* Completed standard chemoradiation with total RT dose of at least 40 Gy and concurrent temozolomide (75mg/m2 daily dose with 80% prescribed dose completed)
* Patients with a tumor that was biopsied or resected in the past followed by observation only without definitive chemoradiation and/or chemotherapy given will be eligible, as long as: repeat maximal surgical resection (biopsy only allowed) has been performed, definitive temozolomide/RT treatment meets the criteria above, and adjuvant temozolomide treatment is planned
* Candidate for adjuvant high dose temozolomide per investigator's clinical judgement
* Adjuvant Temozolomide start date at least 4 weeks, but not more than 6 weeks, from the later of last dose of concomitant temozolomide or radiotherapy
* No evidence of early disease progression per RANO criteria at the time of enrollment
* Women of childbearing potential (WOCBP) must be using a highly effective method of contraception to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug to minimize the risk of pregnancy.

  1. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
  2. Refer to section 10.2.1 for guidance on highly effective contraceptive methods acceptable in this study.
  3. WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as: Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.

Exclusion Criteria:

* Prior treatment with anti-angiogenic agents including bevacizumab.
* Prior treatment with TTFields.
* Progressive disease (according to RANO criteria) after temozolomide/RT.
* Actively participating in another clinical treatment trial intended to treat the underlying astrocytoma.
* Females who are pregnant or breastfeeding.
* Significant co-morbidities at baseline (within 2 weeks prior to adjuvant temozolomide start) which would prevent adjuvant temozolomide treatment:

  1. Thrombocytopenia (platelet count < 100 x 103/μL)
  2. Neutropenia (absolute neutrophil count < 1.5 x 103/μL)
  3. CTC grade 4 non-hematological toxicity (except for alopecia, nausea, vomiting)
  4. Significant liver function impairment - AST or ALT > 5 times the upper limit of normal
  5. Total bilirubin > 2 times upper limit of normal
  6. Significant renal impairment (GFR ≤ 30 ml/min)
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
* A skull defect such as missing bone with no replacement
* Bullet fragments embedded the skull
* Tumors located in the brain stem and/or the cerebellum
* History of hypersensitivity reaction to temozolomide, Dacarbazine (DTIC) or hydrogel.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Tran, MD, PhD, Study Chair — University of Florida
Locations (5):
- United States (5):
  - UF Health at the University of Florida, Gainesville, Florida
  - USF Health Morsani College of Medicine-Moffitt Cancer Center, Tampa, Florida
  - Henry Ford Health System, Detroit, Michigan
  - Brown University-Rhode Island Hospital, Providence, Rhode Island
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Astrocytoma Patients | Control Arm
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled in the control arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Astrocytoma Patients | Control Arm | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Frequency of overall survival in study participants. 2 years of active treatment, lifelong survival follow-up.
Time Frame: Up to 2 years
Population: This multicenter center study was terminated early by mutual decision between the Study Chair/IDE Sponsor and Novocure; therefore, statistical analysis of the 1 participant in the intervention arm was not done.
Arm/Group | Astrocytoma Patients | Control Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: after the start of study treatment for 30 days after the After Treatment Stop Visit
Description: The control arm was a historical control.
Arm/Group | Astrocytoma Patients | Control Arm
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Astrocytoma Patients (N=1) | Control Arm (N=0)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Inpatient Hospitalization for repeat brain tumor resection
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Disease progression
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Astrocytoma Patients (N=1) | Control Arm (N=0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Platelet Count Decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reactive Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
metastatic disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This multicenter center study was terminated early by mutual decision between the Study Chair/IDE Sponsor and Novocure; therefore, statistical analysis of the 1 participant in the intervention arm was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT03906448/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT03906448/ICF_001.pdf